CLINICAL TRIAL: NCT05724914
Title: Clinical Impact in Patients With Delayed Hospitalization in Patients With Out-of-hospital Cardiac Arrest
Brief Title: Call to Door Timing in Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, SungA Bae, Assist Professor, Yonsei University
Other Study IDs: CtD timing
Record Dates: First submitted 2023-01-23; First posted 2023-02-13 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Arrest; Morality
Keywords: Cardiac arrest; Mortality; Timing
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Arrest: Out-Of-Hospital Cardiac Arrest

SUMMARY:
The investigators aimed to investigate the effect of delayed hospitalization on the basis of the call time on the clinical outcomes of patients with OHCA patients using a nationwide OHCA registry.

DETAILED DESCRIPTION:
According to "2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care", immediate call for the local emergency response number takes a key role in the OHCA as the CPR in community does not provide quality of in-hospital CPR. The strong recommendation of speedy transportation, however, does not provide time limitation, and evident data supporting benefit within certain minutes to transfer is lack through our best of search. Therefore, The investigators aimed to investigate the effect of delayed hospitalization on the basis of the call time on the clinical outcomes of patients with OHCA patients using a nationwide OHCA registry.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest event

Exclusion Criteria:

* Arrest of non-cardiac origin
* Age < 18 years
* No any CPR
* Missing data on call time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest with cardiopulmonary resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 182508 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Death from any cause at hospital discharge | up to 30 days
  Death from any cause at hospital discharge

SECONDARY OUTCOMES:
Poor neurological outcomesat hospital discharge | up to 30 days
  poor neurological outcomes, which was defined as a Glasgow-Pittsburge Cerebral Performance Category value at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Yongin Severance Hospital, Yŏngin, Giheung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee OH, Heo SJ, Kim MH, Park JW, Bae S, Kim M, Roh JW, Kim Y, Im E, Jung IH, Cho DK. Therapeutic hypothermia in patients with acute myocardial infarction complicated by out-of-hospital cardiac arrest. BMC Med. 2025 Mar 26;23(1):179. doi: 10.1186/s12916-025-03997-0. PMID 40140891

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT05724914/Prot_SAP_000.pdf